CLINICAL TRIAL: NCT03374696
Title: Prevention of Chlamydia Infection With Theater in School Sex Education - a Randomized Controlled Study
Brief Title: Theater in School Sex Education - a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Annsofie Adolfsson, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Orebro U Sex education
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Attitude; Sexual Behavior; Condom Use; Prevention; Chlamydia Infections; Safe Sex
Keywords: Chlamydia infections; condoms; theater,; sex education
MeSH Terms: conditions — Behavior; Sexual Behavior; Chlamydia Infections; Safe Sex | interventions — Safety

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial with parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention SAFETY was performed in school facilities by professional actors and staff from the municipality's youth guidance center within the county. The actors first enacted a play portraying youths and problems with condom use. Next, a value exercise was held by the youth guidance center staff. The class continued with chlamydia games held by the youth guidance center staff, providing information on symptoms, protection, how to get tested, treatment and consequences. The youth guidance center staff and the actors, playing students, then held a condom school. Lastly, the students came up with new endings to the play. All replays were enacted and the students gave feedback on the new endings. The class ended with condoms being handed out.
  Interventions: Behavioral: SAFETY
- Control group (Active Comparator): The intervention in the control group contained standard education from school staff, based on the sex education guidelines of the Swedish National Agency for Education. Students got education on human sexuality, reproduction, menstruation, love, sex, pregnancy and how STIs and unwanted pregnancy are prevented.
  Interventions: Behavioral: Standard education

INTERVENTIONS:
Behavioral: SAFETY
  Arms: Intervention group
Behavioral: Standard education
  Arms: Control group

SUMMARY:
The study evaluated if interactive theater in school sex education affects student knowledge, attitudes and behavior regarding condom use. The intervention group got a play, value exercises, chlamydia games, condom school and interactive replay with professional actors and staff from a youth guidance center. The control group got standard sex education from school staff, based on the education guidelines of the Swedish National Agency for Education.

DETAILED DESCRIPTION:
The spread of chlamydia indicates that current preventive work with condoms is insufficient. Research shows that reasons behind increased chlamydia include youths taking more sexual risks, due to altered attitudes and sexual behaviors. Since only condoms protect against both sexually transmitted infections (STIs) and unwanted pregnancy, the goal of the World Health Organization (WHO) chlamydia prevention program is to increase condom use. Research suggests that school is the most important arena for sex education, reaching all youths early in life, when many values on sex and relationships are instilled. International studies on theater in sex education indicate effects like increased knowledge on the topic, and partially changed attitudes and behaviors among youths. Furthermore, several studies show that youths feel theater is a good method for sex education and a supplement to standard education.

ELIGIBILITY:
Inclusion Criteria:

* students in eighth grade
* could read and understand Swedish

Exclusion Criteria:

* students in special education.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 826 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
- Knowledge of condom use and chlamydia. - Attitudes toward condom use. - Behavior relating to condom use. | One month.
  Web-based surveys contained questions about
  * knowledge of condom use and chlamydia (7 questions)
  * attitudes toward condom use (5 questions)
  * behavior relating to condom use (6 questions)

CONTACTS AND LOCATIONS:
Overall Officials: Annsofie Adolfsson, Med Dr, Principal Investigator — Orebro University, School of Health Sciences

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary outcome measures will be made available on request.